CLINICAL TRIAL: NCT01431846
Title: Pilot Intervention to Improve the Transition From Hospital to Home
Brief Title: Transition From Hospital to Home Post Cardiac Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RRP 11-242
Record Dates: First submitted 2011-06-23; First posted 2011-09-12 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-09

CONDITIONS: Cardiac Condition
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Discharge Patient (No Intervention): Eight patients who were being discharged from Denver VA Medical Center for cardiac care to their primary care providers were recruited at the time of discharge and completed an interview two weeks following their discharge. Patients were asked to describe their transition to home and identify barriers and facilitators of this process, their understanding of their medical condition, new medications prescribed, timeliness of follow-up visit with their PCP and knowledge of signs/symptoms in which they should seek medical attention.
- Providers (No Intervention): Three providers who refer patients to the Denver VA Medical Center for cardiac care were interviewed to identify barriers and facilitators from their perspective of following-up with patients after their hospitalization at Denver VAMC. Additionally, the same information was asked of providers who participated in two focus groups in the Grand Junction VA.
- Intervention (Experimental): Informed by the interviews and best practices from the literature, pilot test the transitions of care intervention that targets patients and providers to evaluate the feasibility of the intervention to improve process of care measures, including: 1) PCP follow-up within 2-4 weeks of hospital discharge; 2) medications reconciled between pre and post-hospital discharge; 3) discharge summary available to PCP at time of visit; and 4) patient awareness of symptoms that require medical attention
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Informed by the interviews and best practices from the literature, pilot test the transitions of care intervention that targets patients and providers to evaluate the feasibility of the intervention to improve process of care measures, including: 1) PCP follow-up within 2-4 weeks of hospital discharge; 2) medications reconciled between pre and post-hospital discharge; 3) discharge summary available to PCP at time of visit; and 4) patient awareness of symptoms that require medical attention
  Arms: Intervention

SUMMARY:
The study had three parts:

Part 1: Patients (or their home caretakers) who live outside of Denver and receive their primary care at a location other than the Denver VAMC were interviewed after their discharge. The interview covered the patient's perspective about the transition of their medical care from the Denver VA to their primary care facility.

Part 2: Primary care providers from the VA facilities that refer patients to the Denver VA were interviewed regarding their opinions of transition process from the Denver VA back to the primary care VA facilities.

Part 3: The data from the above interviews were used to develop an intervention to improve the transition process from the Denver VA back to the primary care VA facilities.

DETAILED DESCRIPTION:
Aim 1 was to describe barriers and facilitators of the transition process from hospital to home through qualitative interviews among patients discharged from Denver VA Medical Center (tertiary facility) after being transferred from a primary care VA.

Aim 2 was to describe barriers and facilitators of the transition process through qualitative interviews among providers at primary care VA facilities who take care of patients discharged from the Denver VA Medical Center for a cardiac condition.

Aim 3 was to pilot test the transitions of care intervention that targets patients and providers to evaluate the feasibility of the intervention to improve process of care measures, including: 1) PCP follow-up within 2-4 weeks of hospital discharge; 2) medications reconciled between pre and post-hospital discharge; 3) discharge summary available to PCP at time of visit; and 4) patient awareness of symptoms that require medical attention. This pilot was informed by the interviews from Aims 1 and 2 and best practices from the literature. Finally, as part of Aim 3, the primary care providers who saw the patients who completed the pilot were contacted to ask for their input and feedback regarding the pilot project.

Description of Enrolled Population: Study Design and Research Methods This was a mixed methods study where both qualitative and quantitative methods were employed. Through a series of qualitative interviews (n=26), potential barriers and facilitators of the current discharge process were assessed in this hub and spoke model of cardiac care. Informed by these interviews, the transitions of care intervention refined elements from prior studies that have improved this transition process. Finally, a pilot test of this intervention was implemented to assess the effectiveness of the intervention to improve important processes of care during this transition period among patients (n=8) discharged from Denver VAMC after transfer from a primary care VA facility.

ELIGIBILITY:
Inclusion Criteria:

Aims 1 and 3:

* Patients transferred from primary care VA facilities (i.e., Cheyenne, Grand Junction, Sheridan, Ft. Harrison) for cardiac care (e.g., heart failure, acute myocardial infarction) or procedures (coronary angiography, pacemaker implantation) to the Denver VAMC and discharged home to follow-up with their primary care provider, were eligible.

Aim 2:

* Providers from VA primary care facilities, (i.e., Cheyenne, Grand Junction, Sheridan, and Ft. Harrison) who took care of patients discharged from the Denver VAMC for cardiology care, were eligible for the qualitative interviews.

Exclusion Criteria:

Aims 1 and 3:

* Exclusion criteria included:

  * Planned discharge to nursing home or skilled nursing facility;
  * Irreversible, non-cardiac medical condition (e.g. metastatic cancer) likely to affect 6-month survival or ability to execute study protocol;
  * Lack of telephone/ cell phone; and
  * VA is not their primary source of care or their PCP is not in the VA system.

Aim 2: There were exclusion criteria.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ho, MD PhD, Principal Investigator — VA Eastern Colorado Health Care System, Denver, CO
Locations (1):
- VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado, United States

REFERENCES:
- [Result] Hira RS, Kennedy K, Nambi V, Jneid H, Alam M, Basra SS, Ho PM, Deswal A, Ballantyne CM, Petersen LA, Virani SS. Frequency and practice-level variation in inappropriate aspirin use for the primary prevention of cardiovascular disease: insights from the National Cardiovascular Disease Registry's Practice Innovation and Clinical Excellence registry. J Am Coll Cardiol. 2015 Jan 20;65(2):111-21. doi: 10.1016/j.jacc.2014.10.035. PMID 25593051

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Eight patients who were being discharged from Denver VA Medical Center for cardiac care to their primary care providers were recruited at the time of discharge and completed an interview two weeks following their discharge. Patients were asked to describe their transition to home and identify barriers and facilitators of this process, their understanding of their medical condition, new medications prescribed, timeliness of follow-up visit with their PCP and knowledge of signs/symptoms in which they should seek medical attention.
- Arm 2: Three providers who refer patients to the Denver VA Medical Center for cardiac care were interviewed to identify barriers and facilitators from their perspective of following-up with patients after their hospitalization at Denver VAMC. Additionally, the same information was asked of providers who participated in two focus groups in the Grand Junction VA.
- Arm 3: Informed by interviews and best practices from the literature, pilot test the transitions of care intervention that targets patients and providers to evaluate the feasibility of the intervention to improve process of care measures, including: 1)PCP follow-up within 2-4 weeks of hospital discharge; 2) medications reconciled between pre and post-hospital discharge; 3) discharge summary available to PCP at time of visit; and 4) patient awareness of symptoms that require medical attention Intervention: Informed by the interviews and best practices from the literature, pilot test the transitions of care intervention that targets patients and providers to evaluate the feasibility of the intervention to improve process of care measures, including: 1) PCP follow-up within 2-4 weeks of hospital discharge; 2) medications reconciled between pre and post-hospital discharge; 3) discharge summary available to PCP at time of visit; and 4) patient awareness of symptoms that require medical attention
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 8 | 3 | 8
Completed | 8 | 3 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 3: Informed by the interviews and best practices from the literature, pilot test the transitions of care intervention that targets patients and providers to evaluate the feasibility of the intervention to improve process of care measures, including: 1)PCP follow-up within 2-4 weeks of hospital discharge; 2) medications reconciled between pre and post-hospital discharge; 3) discharge summary available to PCP at time of visit; and 4) patient awareness of symptoms that require medical attention
  Intervention: Informed by the interviews and best practices from the literature, pilot test the transitions of care intervention that targets patients and providers to evaluate the feasibility of the intervention to improve process of care measures, including: 1) PCP follow-up within 2-4 weeks of hospital discharge; 2) medications reconciled between pre and post-hospital discharge; 3) discharge summary available to PCP at time of visit; and 4) patient awareness of symptoms that require medical att
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 8 | 3 | 8 | 19
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | NA — provider age not collected | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | 8 | NA — provider age not collected | 8 | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | NA — gender of provider not collected | 4 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 4 | NA — gender of provider not collected | 4 | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: See Primary Outcome Description Below
Description: Follow up appointment within 2 weeks of discharge back to their primary care providers at a primary care facility from a tertiary referral center.
Time Frame: Within 2 weeks of discharge
Measure: Number; unit: participants
Groups:
- Arm 3: Informed by interviews and best practices from the literature, pilot test the transitions of care intervention that targets patients and providers to evaluate the feasibility of the intervention to improve process of care measures, including: 1)PCP follow-up within 2-4 weeks of hospital discharge; 2)medications reconciled between pre and post-hospital discharge; 3)discharge summary available to PCP at time of visit; and 4)patient awareness of symptoms that require medical attention Intervention: Informed by the interviews and best practices from the literature, pilot test the transitions of care intervention that targets patients and providers to evaluate the feasibility of the intervention to improve process of care measures, including: 1) PCP follow-up within 2-4 weeks of hospital discharge; 2) medications reconciled between pre and post-hospital discharge; 3) discharge summary available to PCP at time of visit; and 4) patient awareness of symptoms that require medical attention
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 8 | 3 | 8
participants
  Subjects Interviewed | 8 | 3 | 8
  Follow-up within 2 weeks of discharge | 3 | NA — All providers interviewed to understand facilitators and barriers. This outcome does not pertain to providers. | 6
  Medication reconciliation | 4 | NA — All providers interviewed to understand facilitators and barriers. This outcome does not pertain to providers. | 8
  Discharge Instructions | 8 | NA — All providers interviewed to understand facilitators and barriers. This outcome does not pertain to providers. | 8

ADVERSE EVENTS:
Groups:
- Discharged Patients; Intervention: Total number at risk was 8. Zero adverse events were seen.
- Providers: Total number at risk was 3. Zero adverse events were seen.
Arm/Group | Discharged Patients | Providers | Intervention
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/3 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No